CLINICAL TRIAL: NCT02424383
Title: A Prospective, Multicenter, Single Arm, Real-World Registry Assessing the Clinical Use of the Lutonix 035 Drug Coated Balloon Catheter in Arteries of the Superficial Femoral Artery (SFA) and Popliteal Artery (PA) (SAFE-DCB U.S. Registry)
Brief Title: Real-World Registry Assessing the Clinical Use of the Lutonix 035 Drug Coated Balloon Catheter
Acronym: SAFE-DCB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-14-006
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Diseases; Arterial Occlusive Diseases
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PTA (Lutonix® 035 DCB Catheter) (Experimental): Treatment with the Lutonix 035 DCB will be per the investigational site's standard of care and adhering to the IFU.
  Interventions: Device: PTA (Lutonix® 035 DCB Catheter)

INTERVENTIONS:
Device: PTA (Lutonix® 035 DCB Catheter) — Percutaneous Transluminal Angioplasty (PTA) will involve the insertion of a catheter into one of the femoral arteries. Once the catheter is in place, a tiny balloon on the end of the catheter will be inflated to press against the narrowing (or blockage) in the artery to try to open the blockage, and allow more blood to flow through the artery. The balloon may need to be inflated several times in order for the narrowed area to open up sufficiently to improve the blood flow. The area will be viewed with specialized x-ray or other imaging devices to see if the artery has opened enough.
  The Lutonix® DCB through the blood vessel to the narrowed area to be treated.

SUMMARY:
The objective of this patient registry is to assess the clinical use of the Lutonix 035 DCB PTA Catheter in a heterogeneous patient population in a real world and on-label clinical application.

DETAILED DESCRIPTION:
The registry is a prospective, multicenter, single arm post-market real-world registry in the U.S. assessing the clinical use, safety and outcomes of the Lutonix 035 DCB Catheter in the Superficial Femoral Artery (SFA) and Popliteal Arteries (PA). Registry subjects will be followed for up to three year's post-index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. The subject provides written informed consent using an Informed Consent Form (ICF) that is reviewed and approved by the Institutional Review Board (IRB) for the site.
2. The subject agrees to comply with the protocol-mandated follow-up procedures and visits.
3. The subject is ≥ 21 years old.
4. The subject must have a lesion(s) that can be treated with available Lutonix 035 DCB Catheter according to IFU.

Exclusion Criteria:

1. The subject is unable or unwilling to provide informed consent.
2. The subject is unable or unwilling to comply with the patient registry protocol follow-up procedures and visits.
3. The subject has another medical condition or is currently participating in an investigational drug or an investigational device study that, which, in the opinion of the Investigator, may cause him/her to be non-compliant with the protocol, confounds the data interpretation, or is associated with a life expectancy insufficient to allow for the completion of patient registry procedures and follow-up.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2015-04-23 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2019-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Shammas, MD, Principal Investigator — Midwest Cardiovascular Research Foundation; Edward Woo, MD, Principal Investigator — MedStar Regional
Locations (73):
- United States (73):
  - Lake Martin Laser and Vein Institute, Alexander City, Alabama
  - Chandler Regional Medical Center, Chandler, Arizona
  - St. Luke's Hospital- Phoenix, Phoenix, Arizona
  - UCSD Health System, San Diego, California
  - Colorado Heart and Vascular, Lakewood, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Research Physicians Network Alliance, Boynton Beach, Florida
  - Bradenton Cardiology Center, Bradenton, Florida
  - Clearwater Cardiovascular & Interventional Consultants, Clearwater, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Sarah Cannon Research Institute, LLC, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Orlando Health, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Northside Hospital, Inc, Atlanta, Georgia
  - Vascular Interventional of Thomasville, Associates, Thomasville, Georgia
  - Kaiser Foundation Hospitals, Honolulu, Hawaii
  - Peoria Radiology & Research Foundation, Peoria, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Hutchinson Regional Medical Center - Hutchinson, Inc, Hutchinson, Kansas
  - Maine Medical Center, Portland, Maine
  - MedStar Health Research Institute, Annapolis, Maryland
  - Cape Cod Research Institute, Hyannis, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - DLP Marquette General Hospital, Marquette, Michigan
  - Cardiac & Vascular Research Center of Northern Michigan/McLaren Northern Michigan Hospital, Petoskey, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Merit Health Wesley, Hattiesburg, Mississippi
  - Freeman Health System, Joplin, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cardiovascular Associates of Delaware Valley, Haddon Heights, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - New York Hospital-Queens, Flushing, New York
  - Mount Sinai Beth Israel, New York, New York
  - The Feinstein Institute for Medical Research, New York, New York
  - The Research Foundation for Suny, Syracuse, New York
  - CaroMont Heart Clinical Research, Gastonia, North Carolina
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Carolina East Health System, New Bern, North Carolina
  - Rex Hospital, Inc, Raleigh, North Carolina
  - Mercy West Hospital, Cincinnati, Ohio
  - Jobst Vascular Institute, Toledo, Ohio
  - Jane Phillips Memorial Medical Center, Bartlesville, Oklahoma
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Integris Baptist Medical Center, Inc, Oklahoma City, Oklahoma
  - Providence Health & Service, Portland, Oregon
  - Lankenau Institute for Medical Research, Bryn Mawr, Pennsylvania
  - Saint Vincent Consultants in Cardiovascular Diseases, Erie, Pennsylvania
  - Heart Institute at Largo, Harrisburg, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - The Miriam Hospital - A Lifespan Partner, Providence, Rhode Island
  - Vascular Access Solutions, Orangeburg, South Carolina
  - Stern Cardiovascular Foundation, Inc, Germantown, Tennessee
  - Stern Cardiovascular Foundation Inc., Memphis, Tennessee
  - Seton Heart Institute, Austin, Texas
  - Cardiovascular Specialists of Texas, Austin, Texas
  - Methodist Health System Clinical Research Institute, Dallas, Texas
  - El Paso Cardiology Associates, P.A., El Paso, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Virginia Cardiovascular Specialists, Richmond, Virginia
  - Sentara Medical Group, Virginia Beach, Virginia
  - Lake Washington Vascular, PLLC, Bellevue, Washington
  - CAMC Health Education and Research Institute, Charleston, West Virginia
  - Bellin Memorial Hospital, Inc, Green Bay, Wisconsin
  - Wisconsin Heart-Meriter, Madison, Wisconsin
  - Columbia St. Mary's, Inc., Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 1005 subjects were enrolled and treated with the study device. A total of 966 subjects were included in the Per-Protocol population (excludes subjects with major protocol deviations) for final analysis.
Pre-assignment Details: Between 2015 and 2017, Investigators treated 1005 subjects with the study device. Due to major protocol deviations, 39 subjects were excluded from the analyses conducted in this study. Therefore, the Per-Protocol population included 966 subjects and all outcome results and baseline data are based on this Per-Protocol population.
Groups:
- PTA (Lutonix® 035 DCB Catheter): Treatment with the Lutonix 035 DCB will be per the investigational site's standard of care and adhering to the IFU.
  PTA (Lutonix® 035 DCB Catheter): Percutaneous Transluminal Angioplasty (PTA) will involve the insertion of a catheter into one of the femoral arteries. Once the catheter is in place, a tiny balloon on the end of the catheter will be inflated to press against the narrowing (or blockage) in the artery to try to open the blockage, and allow more blood to flow through the artery. The balloon may need to be inflated several times in order for the narrowed area to open up sufficiently to improve the blood flow. The area will be viewed with specialized x-ray or other imaging devices to see if the artery has opened enough.
  The Lutonix® DCB through the blood vessel to the narrowed area to be treated.
Period: Overall Study
Arm/Group | PTA (Lutonix® 035 DCB Catheter)
Started | 1005
Per-Protocol Population | 966
Completed | 629
Not Completed | 376
Not completed — Withdrawal by Subject | 32
Not completed — Death | 170
Not completed — Sponsor's decision | 3
Not completed — Investigator's decision | 44
Not completed — Lost to Follow-up | 81
Not completed — Other | 7
Not completed — Ineligible for Major Protocol Deviation | 39

BASELINE CHARACTERISTICS:
Population: Only Per-Protocol participants are included in the baseline measures.
Arm/Group | PTA (Lutonix® 035 DCB Catheter)
Number analyzed (Participants) | 966
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age | 69.1 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 418
  Male | 548
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56
  Not Hispanic or Latino | 910
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 192
  White | 735
  More than one race | 0
  Unknown or Not Reported | 20
Region of Enrollment [Number; unit: participants]
  United States | 966
Number of Target Lesions [Number; unit: Participants]
  1 Target Lesion | 744
  2 Target Lesions | 178
  3 Target Lesions | 39
  4 Target Lesions | 5
Number of Devices Used [Number; unit: Participants]
  1 device | 715
  2 devices | 203
  3 devices | 43
  4 devices | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Freedom From Target Lesion Revascularization (TLR) at 12 Months Post Index Procedure
Description: TLR is defined as the first revascularization procedure (e.g. Percutaneous Transluminal Angioplasty (PTA), stenting, etc.) of the target lesion after the index procedure.
Time Frame: 12 months post-index procedure
Population: The number of participants (n) varies from the total number of participants (N) in the study as n depends on the number of participants for which data was available at the given time-point analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTA (Lutonix® 035 DCB Catheter)
Number analyzed (Participants) | 859
percentage of participants | 88.6 [86.3 to 90.6]
Statistical Analysis 1: Comparison: PTA (Lutonix® 035 DCB Catheter); Test type: Other; Freedom from Target LesionRevascularization (TLR) were reported through 12 months with frequency counts, percentages and 95% confidence intervals from exact binomial test. In addition, Kaplan-Meier tables and curves were created

2. Primary Outcome: Percentage of Participants With Freedom From Composite of Device and/or Procedure Related Perioperative Death, Target Limb Major Amputation (Above the Ankle), and Target Vessel Revascularization) at 30 Days Post Index Procedure
Description: Freedom from composite of device and/or procedure related perioperative (≤30 day) death, target limb major amputation (above the ankle), and target vessel revascularization.
Time Frame: 30 days post index procedure
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PTA (Lutonix® 035 DCB Catheter)
Number analyzed (Participants) | 954
Percentage of Participants | 98.2 [97.2 to 98.9]
Statistical Analysis 1: Comparison: PTA (Lutonix® 035 DCB Catheter); Test type: Other; Freedom from composite of safety events from the time following the index procedure through 30 days post procedure were reported with frequency counts, percentages and 95% confidence intervals from exact binomial test. Kaplan-Meier tables and curves were also calculated

3. Secondary Outcome: Percentage of Participants With Freedom From Target Vessel Revascularization (TVR) at 6, 12, 24, and 36 Months Post Index Procedure
Description: TVR is defined as the first revascularization procedure (e.g. Percutaneous Transluminal Angioplasty (PTA), stenting, surgical bypass, etc.) in the target vessel after the index procedure (Kaplan-Meier estimates).
Time Frame: 6 , 12, 24, and 36 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PTA (Lutonix® 035 DCB Catheter)
Number analyzed (Participants) | 966
Percentage of participants
  6 months post index procedure: number analyzed (Participants) | 865
  6 months post index procedure | 94.7 [93.0 to 95.9]
  12 months post index procedure: number analyzed (Participants) | 741
  12 months post index procedure | 86.5 [84.1 to 88.6]
  24 months post index procedure: number analyzed (Participants) | 581
  24 months post index procedure | 75.7 [72.7 to 78.4]
  36 Months Post Index Procedure: number analyzed (Participants) | 223
  36 Months Post Index Procedure | 69.5 [66.2 to 72.6]

4. Secondary Outcome: Percentage of Participants With Freedom From Target Lesion Revascularization (TLR) at 6, 24, and 36 Months Post Index Procedure.
Description: TLR is defined as the first revascularization procedure (e.g. Percutaneous Transluminal Angioplasty (PTA), stenting, etc.) of the target lesion after the index procedure (Kapln-Meier estimates).
Time Frame: 6, 24, and 36 months post index procedure
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PTA (Lutonix® 035 DCB Catheter)
Number analyzed (Participants) | 966
Percentage of Participants
  6 months post index procedure: number analyzed (Participants) | 876
  6 months post index procedure | 95.9 [94.5 to 97.0]
  24 months post index procedure: number analyzed (Participants) | 607
  24 months post index procedure | 79.8 [76.9 to 82.3]
  36 Months Post Index Procedure: number analyzed (Participants) | 240
  36 Months Post Index Procedure | 74.4 [71.2 to 77.2]

5. Secondary Outcome: Percentage of Participants With Acute Device and Procedural Success
Description: Lesion success defined as attainment of < 30% residual stenosis of the target lesion after the index procedure using any percutaneous method and/or non-investigational device (i.e., post-dilatation) and no peri-procedural complications (death, stroke, MI, emergent surgical revascularization, significant distal embolization in target limb, and thrombosis of target vessel) prior to hospital discharge.
Time Frame: At time of Index Procedure
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PTA (Lutonix® 035 DCB Catheter)
Number analyzed (Participants) | 966
Percentage of Participants | 93.0 [91.2 to 94.5]

6. Secondary Outcome: Percentage of Participants With Primary Patency at 12 Months Post Index Procedure
Description: The absence of target lesion restenosis (defined by Duplex Ultrasound (DUS) peak systolic velocity ratio (PSVR) ≥2.5) and freedom from Target Lesion Revascularization (TLR).
  Primary Patency at 12-Months post index-procedure by Kaplan-Meier estimates using a Method in which all subjects without a confirmed TLR or loss of patency were censored at Day 395 or the date of study discontinuation, whichever occurred first.
Time Frame: 12 months post-index procedure
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PTA (Lutonix® 035 DCB Catheter)
Number analyzed (Participants) | 714
Percentage of Participants | 83.7 [81.1 to 86.0]

7. Secondary Outcome: Percentage of Participants With Freedom From Composite of All-cause Perioperative (≤30 Day) Death and From the Following: Index Limb Amputation, Index Limb Reintervention, and Index-limb-related Death at 6, 12, 24, and 36 Months Post Index Procedure
Description: Freedom from composite of all-cause perioperative (≤30 day) death and from the following: index limb amputation, index limb reintervention, and index-limb-related death (Kaplan-Meier estimates).
Time Frame: 6, 12, 24, and 36 Months Post Index Procedure
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PTA (Lutonix® 035 DCB Catheter)
Number analyzed (Participants) | 966
Percentage of Participants
  6 months post index procedure: number analyzed (Participants) | 930
  6 months post index procedure | 90.3 [88.2 to 92.1]
  12 months post index procedure: number analyzed (Participants) | 884
  12 months post index procedure | 80.8 [78.0 to 83.3]
  24 months post index procedure: number analyzed (Participants) | 820
  24 months post index procedure | 67.4 [64.1 to 70.6]
  36 Months Post Index Procedure: number analyzed (Participants) | 762
  36 Months Post Index Procedure | 58.4 [54.8 to 61.9]

8. Secondary Outcome: Percentage of Participants With Freedom From Major Amputation of the Target Limb (Above the Ankle Amputation) at 6, 12, 24, and 36 Months Post Index Procedure.
Description: Freedom from major amputation of the target limb defined as above the ankle amputation
Time Frame: 6, 12, 24, and 36 Months Post Index Procedure
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PTA (Lutonix® 035 DCB Catheter)
Number analyzed (Participants) | 966
Percentage of Participants
  6 months post index procedure: number analyzed (Participants) | 916
  6 months post index procedure | 98.5 [97.4 to 99.2]
  12 months post index procedure: number analyzed (Participants) | 857
  12 months post index procedure | 97.5 [96.3 to 98.5]
  24 months post index procedure: number analyzed (Participants) | 772
  24 months post index procedure | 96.6 [95.1 to 97.8]
  36 Months post Index Procedure: number analyzed (Participants) | 682
  36 Months post Index Procedure | 95.6 [93.8 to 97.0]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from the index procedure through final contact with the participants (36 months post index procedure), or early termination and include events experienced by ALL enrolled participants (1005).
Arm/Group | PTA (Lutonix® 035 DCB Catheter)
All-Cause Mortality (participants affected / at risk) | 173/1005
Serious Adverse Events (participants affected / at risk) | 65/1005
Other Adverse Events (participants affected / at risk) | 121/1005
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTA (Lutonix® 035 DCB Catheter) (N=1005)
Atrial Fibrillation (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 3
Vessel Puncture Site Haematoma (General disorders) | 4
Complication of Device removal (General disorders) | 1
Impaired Healing (General disorders) | 1
Thrombosis in Device (General disorders) | 1
Contrast Media Allergy (Immune system disorders) | 1
Gangrene (Infections and infestations) | 1
Vessel Puncture Site Infection (Infections and infestations) | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 8
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 5
Procedural Complication (Injury, poisoning and procedural complications) | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1
Peripheral Artery Dissection (Vascular disorders) | 25
Peripheral Arterial Occlusive Disease (Vascular disorders) | 7
Vessel Perforation (Vascular disorders) | 4
Embolism Arterial (Vascular disorders) | 2
Peripheral Artery Stenosis (Vascular disorders) | 2
Peripheral Artery Thrombosis (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Vasospasm (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTA (Lutonix® 035 DCB Catheter) (N=1005)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Retroperitoneal Hemorrhage (Gastrointestinal disorders) | 3 (3)
Vessel Puncture Site Hematoma (General disorders) | 18 (18)
Local Swelling (General disorders) | 4 (4)
Vessel Puncture Site Hemorrhage (General disorders) | 2 (2)
Vessel Puncture Site swelling (General disorders) | 2 (2)
Complication of Device Removal (General disorders) | 1 (1)
Thrombosis in device (General disorders) | 1 (1)
Vessel Puncture Site Pain (General disorders) | 1 (1)
Contrast Media Allergy (Immune system disorders) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Vessel Puncture Site Infection (Infections and infestations) | 1 (1)
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 13 (13)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 10 (11)
Procedural Complication (Injury, poisoning and procedural complications) | 3 (3)
Procedural Pain (Injury, poisoning and procedural complications) | 3 (3)
Scrotal Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral Artery Dissection (Vascular disorders) | 32 (32)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 7 (7)
Vessel Perforation (Vascular disorders) | 5 (5)
Peripheral Artery Stenosis (Vascular disorders) | 4 (4)
Peripheral Artery Thrombosis (Vascular disorders) | 4 (4)
Embolism Arterial (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 3 (3)
Arteriovenous Fistula (Vascular disorders) | 2 (2)
Vasospasm (Vascular disorders) | 2 (2)
Peripheral Artery Aneurysm (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT02424383/Prot_SAP_000.pdf